CLINICAL TRIAL: NCT04080531
Title: Influenza Vaccination in Plasma Cell Dyscrasias
Brief Title: Influenza Vaccination for Flu Prevention in Patients With Plasma Cell Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry); National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig Hofmeister, Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00111721; NCI-2019-03734 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship4709-19 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2019-09-04; First posted 2019-09-06 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Plasma Cell Neoplasm
MeSH Terms: conditions — Neoplasms, Plasma Cell | interventions — 13-valent pneumococcal vaccine; Influenza Vaccines; Fluzone High-Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (trivalent influenza vaccine, Prevnar) (Experimental): Patients receive trivalent influenza vaccine IM at weeks 1, 9, and 17, and pneumococcal 13-valent conjugate vaccine IM at week 5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Trivalent Influenza Vaccine
- Arm II (trivalent influenza vaccine, Prevnar) (Experimental): Patients receive trivalent influenza vaccine IM at week 1 and pneumococcal 13-valent conjugate vaccine IM at week 5 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Trivalent Influenza Vaccine

INTERVENTIONS:
Biological: Pneumococcal 13-valent Conjugate Vaccine — Given IM
  Other Names: PCV13; Prevnar 13
Biological: Trivalent Influenza Vaccine — Given IM
  Other Names: Flu shot; Flu vaccination; Fluzone; Fluzone HD; Fluzone High-dose; Influenza Vaccine; Influenza Virus Vaccine, Trivalent, Types A and B; TIV

SUMMARY:
This phase IV trial studies how well influenza vaccination works in preventing infections such as influenza in patients with plasma cell disorders. Influenza infections may theoretically support the growth of tumor cells and improving protection against influenza may improve the status of patients' plasma cell disorder. Giving influenza vaccination may reduce influenza-related complications including infections, hospitalizations, and deaths, and improve the status of plasma cell disorders.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Demonstrate an absolute 25% increase in seroprotection, defined as hemagglutination antibody inhibition (HAI) > 40 against all strains, at week 21 in the experimental arm compared to the control arm.

II. Determine correlation between HAI, predefined risk of influenza-like illness (low, moderate, high), and progression-free survival (PFS).

EXPLORATORY OBJECTIVES:

I. Measurement of B & T-cell subsets and flu-specific responses as a way of understanding immunosuppression in this patient population, correlating with influenza-like illness.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive trivalent influenza vaccine intramuscularly (IM) at weeks 1, 9, and 17, and pneumococcal 13-valent conjugate vaccine IM at week 5 in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive trivalent influenza vaccine IM at week 1 and pneumococcal 13-valent conjugate vaccine IM at week 5 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed for 4 weeks and then periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a plasma cell dyscrasia that fits in the International Myeloma Working Group (IMWG) diagnostic criteria.
* Both men and women of all races and ethnic groups are eligible for this study.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3 (Karnofsky ≥ 30%) is required for eligibility.
* Patient must be eligible to receive standard of care influenza vaccination. If the patient has a history of egg allergy with symptoms more severe than urticaria, e.g. angioedema, respiratory distress, lightheadedness, or recurrent emesis, they remain eligible to receive influenza vaccination but must receive the vaccine in a facility able to recognize and manage severe allergic reactions. Persons who are able to eat lightly cooked egg (e.g., scrambled egg) without reaction are unlikely to be allergic, although egg-allergic persons might tolerate egg in baked products.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have already received the seasonal influenza vaccine in the current season.
* History of Guillain-Barré syndrome.
* Patients with a previous severe allergic reaction to influenza vaccination or pneumococcal 13-valent conjugate vaccine (PCV13).
* Expected survival < 9 months.
* Prisoners.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-05-11 (Actual); Study Completion 2022-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Hofmeister, MD, MPH, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Trivalent Influenza Vaccine, Prevnar) | Arm II (Trivalent Influenza Vaccine, Prevnar)
Started | 80 | 85
Completed | 64 | 81
Not Completed | 16 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Trivalent Influenza Vaccine, Prevnar) | Arm II (Trivalent Influenza Vaccine, Prevnar) | Total
Number analyzed (Participants) | 80 | 85 | 165
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 47 | 93
  >=65 years | 34 | 38 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.7 (11.60) | 62.8 (9.68) | 62.35 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 30 | 67
  Male | 43 | 55 | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 70 | 83 | 153
  Unknown or Not Reported | 8 | 1 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 22 | 27 | 49
  White | 51 | 54 | 105
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 80 | 85 | 165

OUTCOME MEASURES:

1. Primary Outcome: Seroprotection Based on Hemagglutination Antibody Inhibition (HAI)
Description: HAI in blood at week 21 for all variants
Time Frame: 21 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Trivalent Influenza Vaccine, Prevnar) | Arm II (Trivalent Influenza Vaccine, Prevnar)
Number analyzed (Participants) | 80 | 85
Participants | 32 | 22

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm I (Trivalent Influenza Vaccine, Prevnar) | Arm II (Trivalent Influenza Vaccine, Prevnar)
All-Cause Mortality (participants affected / at risk) | 3/80 | 1/85
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/85
Other Adverse Events (participants affected / at risk) | 0/80 | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT04080531/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT04080531/ICF_002.pdf